CLINICAL TRIAL: NCT04287569
Title: Use of Multispectral Imaging in Digestive Inflammation Diagnosis
Brief Title: Multispectral Imaging Endoscopy in Digestive Inflammation
Acronym: ENDOSPECTRALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P160409J; 2019-A01602-55 (Registry Identifier: IDRCB)
Record Dates: First submitted 2019-12-16; First posted 2020-02-27 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2022-04

CONDITIONS: Digestive Inflammation
Keywords: digestive inflammation; multispectral imaging; multispectral gastroscopy; multispectral coloscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- video recording of endoscopy (Experimental): Record of sequences of video-endoscopy and the reflectance of light through fibroscopy
  Interventions: Device: Record during endoscopy of video-endoscopy sequences and reflectance

INTERVENTIONS:
Device: Record during endoscopy of video-endoscopy sequences and reflectance — Record of video-endoscopy sequences and reflectance, during endoscopy with biopsy.

SUMMARY:
The study aims as principal objective to show the association between reflectance intensity of mucosa at different wave lengths and

* the presence of acute or chronic inflammation in stomach or rectum and normal mucosa;
* the presence of glandular atrophy in stomach or intestinal metaplasia.

The secondary objectives are:

* to identify reflectance profile which characterize an acute or a chronic inflammation, a glandular atrophy or an intestinal metaplasia, respectively;
* to find a correlation between the reflectance to different frequencies and intensity of inflammation according to Sydney Classification in stomach (Dixon M F 1994) and in rectum (Erben U 2014).

DETAILED DESCRIPTION:
This is a comparative, prospective, non randomized, controled, mono-centric study.

Eligible patients: patients planned to undergo an upper gastrointestinal endoscopy or a rectosigmoidoscopy with biopsy in the digestive endoscopy unit of Hôpital Ambroise Paré. For patients accept participating to the study and sign the informed consent, they will be enrolled in the study and the recorded imaging of stomach or rectum will be obtained.

Patient management will not be modified in this study as compared to usual endoscopy procedure. Multispectral endoscopy will only prolong the examination 1 minute in order to obtain the imaging. The study consists of video records of endoscopy with white light and the reflected light projected by the fibre introduced 60 seconds in examined channel. This reflected light will be redirected to a multispectral camera.

The endoscopy examinations will be performed in gastric antrum and cardia when theses sites present abnormal position or contour. The biopsies samples of gastric mucosa will be performed in the antrum or the cardia according to the Guideline of the Société Française d'Endoscopie Digestive.

6 groups of patients will be constituted (included 2 groups of control) as described below and compared posteriorly:

* The control group of rectum: 20 patients with negative result of endoscopy examination (-) and negative result of anatomopathological analysis (-);
* The group of 20 patients with positive result of endoscopy examination (+) and positive result of anatomopathological analysis (+) in rectum;
* The group of 20 patients with negative result of endoscopy examination (-) and positive result of anatomopathological analysis (+) in rectum;
* The control group of stomach: 60 patients with negative result of endoscopy examination (-) and negative result in anatomopathological analysis (-);
* The group of 45 patients with positive result of endoscopy examination (+) and positive result of anatomopathological analysis (+) in stomach;
* The group of 30 patients with negative result of endoscopy examination (-) and positive result of anatomopathological analysis (+) in stomach.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing a digestive endoscopy under general anesthesia, or a rectoscopy without anesthesia, with indicators of systematic biopsy regardless of reason;
* Aged ≥ 18 years;
* Covered by a public health insurance regime;
* Signed consent.

Exclusion Criteria:

* History of gastric or rectal surgery regardless of nature;
* Gastrointestinal bleeding by hematemesis or rectal bleeding;
* Hemostasis disorders preventing biopsy.
* Difficulties in understanding french language;
* Pregnant or breast feeding woman;
* Woman of childbearing age without reliable contraception;
* Adult under legal protection with tutor or curator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Reflectance endoscopy for gastric mucosa with lesions | Up to 12 months
  The reflectance endoscopy for gastric and rectal mucosa in different wavelength of presence of the lesions, in comparison with anatomopathological analysis on gastric and rectal mucosa, to diagnosis acute and chronic inflammation, glandular atrophy and intestinal metaplasia.
  This outcome will show reflectance for mucosa in presence of lesions which classified by anatomopathological analysis: comparison report.

SECONDARY OUTCOMES:
Statistic association between profiles of reflectance and anatomopathological classifications | Up to 12 months
  Statistic association between the profiles of reflectance in different frequencies and anatomopathological classifications in stomach and rectal analysis (such as acute or chronic inflammation, glandular atrophy and intestinal metaplasia).
Correlation between reflectance and intensity of inflammation | Up to 12 months
  Correlation between reflectance to different frequencies and intensity of inflammation in stomach (according to the Classification of Sydney) and in rectum (according to Erben et al).
Sub-study: morphological comparison between 2D/3D reconstruction and endoscopist's description | Up to 12 months
  Morphological comparison between reconstruction in 2D or 3D and morphological description of mucosa (the antra and the cardia) by endoscopist.
  The type of method as structure from motion (SFM) should be used to map in 3D or 2D the antra, few publication show method of mapping in 3D or 2D for hollow organs, potentially transformable and utilisable under clinical condition.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Lamarque, MD, PhD, Principal Investigator — Service Hépato-Gastroentérologie, Hôpital Ambroise Paré, Boulogne Billancourt
Locations (1):
- Service Hépato-Gastroentérologie, Hôpital Ambroise Paré, Boulogne-Billancourt, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No